CLINICAL TRIAL: NCT03193801
Title: PARTNER 3 Trial - SAPIEN 3 Transcatheter Heart Valve Implantation in Patients With a Failing Mitral Bioprosthetic Valve
Brief Title: PARTNER 3 Trial - Mitral Valve in Valve
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-08 MVIV
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Disease; Mitral Valve Regurgitation; Heart Failure
Keywords: SAPIEN 3; PARTNER 3; cardiovascular disease; TMVR; failing valve; failing bioprosthetic valve
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Failing mitral transcatheter valve (Experimental): Patients with a failing bioprosthetic valve in the mitral position demonstrating stenosis and/or insufficiency will be treated with Edwards SAPIEN 3 transcatheter valve.
  Interventions: Device: Edwards SAPIEN 3 transcatheter valve, Model 9600TFX

INTERVENTIONS:
Device: Edwards SAPIEN 3 transcatheter valve, Model 9600TFX — Edwards SAPIEN 3 THV system Model 9600TFX with the associated delivery systems.
  Other Names: TMVR

SUMMARY:
To assess the safety and effectiveness of the SAPIEN 3 transcatheter heart valve in patients with a failing mitral bioprosthetic valve.

DETAILED DESCRIPTION:
A prospective, single-arm, multicenter clinical trial. This study will enroll patients with symptomatic heart disease due to a failing bioprosthetic mitral valve (stenosed, insufficient, or combined).

ELIGIBILITY:
Inclusion Criteria:

1. Failing surgically implanted bioprosthetic valve in the mitral position demonstrating ≥ moderate stenosis and/or ≥ moderate insufficiency.
2. Surgical bioprosthetic valve with a true internal diameter (True ID) of 16.5 mm to 28.5 mm.
3. NYHA Functional Class ≥ II.
4. Heart Team agrees the patient is intermediate risk (i.e. STS score of ≥3 and < 8).
5. Heart Team agrees valve implantation will likely benefit the patient.
6. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) / Ethics Committee (EC) of the respective clinical site.

Exclusion Criteria:

1. Index valve has ≥ mild paravalvular regurgitation where the surgical bioprosthesis is not securely fixed in the native annulus or is not structurally intact as determined by transesophageal echocardiography (TEE).
2. Surgical or transcatheter aortic valve placed so that extension into left ventricular outflow tract (LVOT) that may impinge on the mitral implant.
3. Known residual mean gradient >10 mmHg at the end of the index procedure for implantation of the original surgical valve.
4. Severe right ventricle (RV) dysfunction.
5. Anatomical characteristics that would preclude safe access to the apex (transapical).
6. Severe regurgitation or stenosis of any other valve.
7. Severe lung disease (FEV1 < 50% predicted) or currently on home oxygen
8. Severe pulmonary hypertension (e.g., PA systolic pressure ≥ 2/3 systemic pressure)
9. Anatomical characteristics that would increase risk of LVOT obstruction (e.g., aortomitral angle, LVOT size, etc.).
10. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before enrollment.
11. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days prior to the index procedure. Implantation of a permanent pacemaker (PPM) or implantable cardioverter defibrillator (ICD) is not considered an exclusion.
12. Patients with planned concomitant surgical or transcatheter ablation for atrial fibrillation.
13. Leukopenia (white blood count < 3000 cell/mL), anemia (hemoglobin < 9 g/dL), thrombocytopenia (blood platelet count < 50,000 cell/mL), history of bleeding diathesis or coagulopathy, or hypercoagulable states.
14. Untreated clinically significant coronary artery disease requiring revascularization.
15. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation, or mechanical heart assistance within 30 days of enrollment.
16. Emergency intervention/surgical procedures within one month (30 days) prior to the procedure.
17. Any planned surgical, percutaneous coronary, or peripheral procedure to be performed within the 30-day follow-up from the procedure.
18. Hypertrophic cardiomyopathy with obstruction (HOCM).
19. Left ventricular ejection fraction (LVEF) < 30%.
20. Cardiac imaging evidence of intracardiac mass, thrombus, or vegetation.
21. Inability to tolerate or condition precluding treatment with antithrombotic/anticoagulation therapy during or after the valve implant procedure.
22. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with premedication.
23. Stroke or transient ischemic attack (TIA) within 90 days of enrollment.
24. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of enrollment.
25. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy at the time of screening.
26. Active bacterial endocarditis within 6 months (180 days) of the procedure.
27. Patient refuses blood products.
28. Estimated life expectancy < 24 months.
29. Currently participating in an investigational drug or another device study. Note: Clinical trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
30. Positive urine or serum pregnancy test in female subjects of childbearing potential.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2031-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mayra Guerrero, MD, Principal Investigator — Mayo Clinic; Chris S. Malaisrie, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Alan Zajarias, MD, Principal Investigator — Washington University School of Medicine
Locations (12):
- United States (9):
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northshore University Health System Research Institution, Evanston, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital/ Washington University, St Louis, Missouri
  - NYU Lagone Medical Center, New York, New York
  - Providence Heart & Vascular Institution, Portland, Oregon
  - The Heart Hospital of Baylor Plano, Plano, Texas
- The Prince Charles Hospital, Chermside, Queensland, Australia
- Brazil (2):
  - Instituto do Coração da Universidade de São Paulo, Cerqueira César, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, Vila Mariana, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malaisrie SC, Guerrero M, Davidson C, Williams M, de Brito FS Jr, Abizaid A, Shah P, Kaneko T, Poon K, Levisay J, Yu X, Pibarot P, Hahn RT, Blanke P, Leon MB, Mack MJ, Zajarias A; PARTNER 3 Mitral Valve-in-Valve Study Investigators. One-Year Outcomes of Transseptal Mitral Valve-in-Valve in Intermediate Surgical Risk Patients. Circ Cardiovasc Interv. 2024 Aug;17(8):e013782. doi: 10.1161/CIRCINTERVENTIONS.123.013782. Epub 2024 Jul 22. PMID 39034924

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Failing Mitral Transcatheter Valve
Started | 53
Completed | 50
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Failing Mitral Transcatheter Valve
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black or African American | 4
  White | 31
  Other | 7
  Unknown | 5
Region of Enrollment [Number; unit: participants]
  United States | 34
  Brazil | 12
  Australia | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety and Effectiveness - Composite of All-cause Mortality and Stroke
Description: Non-hierarchical composite endpoint of all-cause mortality and stroke at 1-year post-procedure
Time Frame: 1 Year
Population: Valve implant population
Measure: Count of Participants; unit: Participants
Arm/Group | Failing Mitral Transcatheter Valve
Number analyzed (Participants) | 50
Participants | 0

2. Secondary Outcome: New York Heart Association (NYHA) Functional Class - Change From Baseline
Description: NYHA is a functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort.
  A decrease in NYHA class (negative value) shows patient improvement at 30 days.
Time Frame: 30 Days
Population: Valve implant population - 2 subjects did not complete the 30-day visit.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Failing Mitral Transcatheter Valve
Number analyzed (Participants) | 48
score on a scale | -1.4 (0.73)

3. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) - Change From Baseline
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom, social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  An increase in KCCQ score (positive value) shows patient improvement at 30 days.
Time Frame: 30 days
Population: Valve implant population - 2 subjects did not complete the 30-day visit.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Failing Mitral Transcatheter Valve
Number analyzed (Participants) | 48
score on a scale | 31.0 (26.06)

4. Secondary Outcome: Mitral Regurgitation - Change From Baseline
Description: Echocardiographic assessment of the degree of mitral valve regurgitation
  None=0, Trace=0.5, Mild or Mild-Moderate=1, Moderate=2, Moderate-Severe=3, and Severe=4.
  A decrease in MR (negative value) shows patient improvement at 30 days.
Time Frame: 30 days
Population: Valve implant population - 4 subjects did not receive an echocardiogram at 30 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Failing Mitral Transcatheter Valve
Number analyzed (Participants) | 46
score on a scale | -1.4 (1.48)

5. Secondary Outcome: Pulmonary Artery Systolic Pressure - Change From Baseline
Description: Echocardiographic assessment of pulmonary artery systolic pressure
  A decrease in pulmonary artery systolic pressure (negative value) shows patient improvement at 30 days.
Time Frame: 30 days
Population: Valve implant population - 35 subjects had data at 30 days
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Failing Mitral Transcatheter Valve
Number analyzed (Participants) | 35
mmHg | -9.5 (14.64)

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Failing Mitral Transcatheter Valve
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 21/50
Other Adverse Events (participants affected / at risk) | 15/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Failing Mitral Transcatheter Valve (N=50)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Myelitis (Infections and infestations) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Vascular pseudoaneurysm thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Transvalvular pressure gradient increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Device deployment issue (Product Issues) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Failing Mitral Transcatheter Valve (N=50)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 3 (3)
Prosthetic cardiac valve stenosis (General disorders) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03193801/Prot_SAP_000.pdf